CLINICAL TRIAL: NCT02485821
Title: Vaginal Estradiol Pretreatment in Labour Induction With Misoprostol
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Mohamed S. Sweed lecturer of Obstetrics & Gynecology AinShams University., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS39825273
Record Dates: First submitted 2015-06-19; First posted 2015-06-30 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Failed Induction of Labor
Keywords: Estradiol; Misoprostol; Induction of labor; Cervical ripening; Bishop score
MeSH Terms: interventions — Estradiol; Ethinyl Estradiol; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Estradiol + Misoprostol (Experimental): 100 patient will receive single dose vaginal estradiol 50mcg tablet (Ethinyl Estradiol manufactured by KAHIRA Pharmaceutical company) and vaginal misoprostol 25mcg tablet (Vagiprost manufactured by ADWIA Pharmaceutical company), misoprostol alone will repeated every 6hours up to five doses.
  Interventions: Drug: Estradiol; Drug: Misoprostol
- Placebo + Misoprostol (Placebo Comparator): 100 patients will receive placebo vaginally and misoprostol 25 mcg which will be repeated every 6 hours up to five doses.
  Interventions: Drug: Placebo; Drug: Misoprostol

INTERVENTIONS:
Drug: Estradiol
  Other Names: Ethinyl Estradiol
  Arms: Estradiol + Misoprostol
Drug: Placebo
  Arms: Placebo + Misoprostol
Drug: Misoprostol
  Other Names: Vagiprost

SUMMARY:
To assess the effect of vaginal estradiol pretreatment before vaginal misoprostol on labor induction.

DETAILED DESCRIPTION:
A prospective double blind randomized clinical trial. Conducted at Ain Shams University Maternity Hospital. Patients fulfilling inclusion and exclusion criteria will be divided into two groups. Group (A):

100 patient will receive single dose vaginal estradiol 50mcg tablet (Ethinyl Estradiol manufactured by KAHIRA Pharmaceutical company) and vaginal misoprostol 25mcg tablet (Vagiprost manufactured by ADWIA Pharmaceutical company), misoprostol alone will repeated every 6hours up to five doses.

Group (B):

100 patients will receive placebo vaginally and misoprostol 25 mcg which will be repeated every 6 hours up to five doses.

Primary Outcome

* Measure the time to cervical ripening. Secondary Outcome
* Measure the time to active labor.
* Number of misoprostol doses.
* Induction delivery time.
* Time to achieve vaginal delivery.
* Fetal outcome (Apgar score).

ELIGIBILITY:
Inclusion criteria:

* Maternal age ≥ 18 years old.
* Gestational age ≥ 37 wks to 41 wks.
* BMI between 20 kg/m2 and 35kg/m2.
* Vertex presentation.
* Singleton pregnancy.

Exclusion criteria:

* Multiple pregnancy.
* Non vertex presentation.
* Absolute or relative contraindication to vaginal delivery e.g. (Placenta previa, fibroid uterus, uterine anomalies, previous uterine surgery).
* PROM.
* IUFD.
* Fetal distress.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Time to cervical ripening. | 24 hours

SECONDARY OUTCOMES:
Time to active labor | 30 hours
Number of misoprostol doses | 24 hours
Induction delivery time | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Osama El-Kady, MD, Principal Investigator — AinShams University; AbdEl-Latif El-Kholy, MD, Principal Investigator — AinShams University
Locations (1):
- Ain Shams University, Cairo, Egypt